CLINICAL TRIAL: NCT05254691
Title: Measuring Work-of-Breathing in Mechanically Ventilated Children
Brief Title: WOB and Paediatric Mechanical Ventilation
Acronym: PedWOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Martin Kneyber, MD PhD FCCM, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL38361.042.11
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Pediatric Respiratory Diseases; Ventilator Weaning; Respiration, Artificial; Respiratory Failure; Pediatrics; Work of Breathing
Keywords: pediatrics; mechanical ventilation; work of breathing
MeSH Terms: conditions — Respiratory Aspiration; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: This is a prospective exploratory study with invasive measurements in a 20 bed tertiary paediatric intensive care facility at the Beatrix Children's Hospital/University Medical Centre Groningen.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): All children are put on a time-cycled, pressure limited ventilation mode (AVEA, CareFusion, Yorba Linda, CA, USA). Inspiratory pressures are set to deliver a expiratory tidal volume of 5-7 ml/kg ideal bodyweight. The frequency of the delivered machine-breaths is set in accordance with age and disease condition of the patient. Then the patient set rate of breaths per minute delivered by the ventilator is reduced with 25%, allowing for more spontaneous breaths.
- Sprinting (Experimental): The ventilator mode is switched to PS ventilation. The level of PS is set to meet the level of PS set when the patient is ventilated in the SIMV-PS mode. The patient will be in the PS mode until he or she clinically shows increased work-of-breathing (tachypnoea and the presence of nasal flaring and intercostal and/or interjugular retractions indicate increased work of breathing).
  Interventions: Procedure: Sprinting

INTERVENTIONS:
Procedure: Sprinting — The ventilator mode is switched to PS ventilation. The level of PS is set to meet the level of PS set when the patient is ventilated in the SIMV-PS mode. The patient will be in the PS mode until he or she clinically shows increased work-of-breathing (tachypnoea and the presence of nasal flaring and intercostal and/or interjugular retractions indicate increased work of breathing). This "sprinting" is performed on the theory that the respiratory muscles can be slowly trained to sustain complete spontaneous breathing. Also, theoretically this "sprinting" allows a better global and regional distribution of the tidal volume in the lung.
  Arms: Sprinting

SUMMARY:
Rationale: The most common approach to weaning infants and children is gradual reduction of ventilatory support ("traditional approach"). Alternatively, another approach to weaning is attempted with alternating periods of complete ventilatory support and graded spontaneous breathing with assistance ("sprinting approach"). Both approaches are used randomly in our unit: the decision to use which approach is dependent upon the preferences of the attending physician as described in many observational single center studies. To date, there is no data comparing the safety and efficacy of the "sprinting" approach with more traditional approaches of weaning in children. Hence, numerous issues remain unanswered, including the work-of-breathing during each approach. For this research proposal, we want to measure the work-of-breathing daily, using the traditional approach (the area under the oesophageal pressure - volume curve) and study its correlation with clinical parameters and EMG activity of the diaphragm and intercostal muscles from the moment that the patient is weaned off the ventilator.

Objective: The primary objective for this study is to compare for each patient of the work-of-breathing during the "sprinting"approach and the "traditional approach.The secondary objectives for this study are to compare the oesophageal pressure rate and (PRP) and pressure time product (PTP), the PaO2/FiO2 ratio, global and regional distribution of tidal volume measured using electrical impedance tomography (EIT), phase distribution of the respiratory inductive plethysmography (RIP) signal and the EMG activity of the diaphragm and intercostal muscles between the "sprinting"and the "traditional" approach..

Study design: This is a prospective exploratory study with invasive measurements in a 20 bed tertiary paediatric intensive care facility at the Beatrix Children's Hospital/University Medical Centre Groningen.

Study population: All mechanically ventilated children aged 0 to 5 years with or without lung pathology admitted to the paediatric intensive care unit are eligible for inclusion. Inclusion criteria include mechanical ventilation for at least 48 hours, weight ≥ 3 kg, sufficient respiratory drive present, deemed eligible for weaning by the attending physician, and stable haemodynamics (defined by the absence of need for increase in vaso-active drugs and/or fluid challenges at least 6 hours prior to enrolment). Exclusion criteria include mechanical ventilation less than 48 hours, not eligible for weaning (usually when there are unstable ventilator settings, defined by the need for increase of inspiratory pressures or positive end-expiratory pressure, and a FiO2 > 0.6 within 6 hours prior to enrolment), unstable haemodynamics (defined by the need for increase in vaso-ative drugs and/or fluid challenges within 6 hours prior to enrolment), leakage around the endotracheal tube > 5%, admitted to the neonatal intensive care unit, preterm birth with gestational age corrected for post-conceptional age less than 40 weeks, congenital or acquired neuromuscular disorders, congenital or acquired central nervous system disorders with depressed respiratory drive, congenital or acquired damage to the phrenic nerve, congenital or acquired paralysis of the diaphragm, use of neuromuscular blockade prior to enrolment, uncorrected congenital heart disorder, and chronic lung disease.

Main study parameters/endpoints: The main study parameter is the level and time course of the patient's work-of-breathing mathematically calculated by the area under the pressure-volume curve Secondary study parameters include the level and time course of the PRP and PTP, level and time course of oxygenation (PaO2/FiO2 ratio), global and regional distribution of tidal volume, phase distribution, EMG activity of the diaphragm and intercostal muscles, heart rate, respiratory rate..

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are a priori no specific benefits for the patients who participate in the study.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE The need for mechanical ventilation for respiratory failure is one the most common indications for children to be admitted to a centralized paediatric intensive care unit (PICU) in the Netherlands. Up to 64% of all admitted children need mechanical ventilation for at least 24 hrs (1,2). Hence mechanical ventilation is a key feature in the management of critically ill children. Nevertheless, numerous issues related to the use of mechanical ventilation in children remain unsolved. Much of the current clinical practice is based upon anecdotal experience and data obtained from studies performed in critically ill adults (3). However, the respiratory system is physiologically different between small babies, children and adults implying that all data obtained from adults cannot be easily extrapolated to children (4). For instance (to name but a few), the elastic properties of the lung increases during childhood contributing to increased lung compliance. Furthermore, over the remainder of childhood the lung continues to grow and mature: at the age of 8 years the alveolar surface is about half of that of an adult. Interalveolar pores develop during pre-school years, whereas broncho-alveolar pores begin to develop at the age of 6 - 8 years. The absence of these collateral pathways places children at risk for the development of atelectasis and resulting ventilation/perfusion inequality. Next to this, the resistance of peripheral airways decreases profoundly with increasing age. However, the resistance in an 8-year old is still four times higher than in an adult. Tidal volume (Vt) is comparable between children and adults (about 5 - 7 ml/kg ideal bodyweight), but functional residual capacitity (FRC) in young children is much smaller than in adults. And finally, chest wall compliance is also profoundly different between young children and adults. The chest wall compliance decreases with increasing age because of ossification of the rib cage and an increase in mucular tone of the intercostal muscles.

   Although mechanical ventilation is often life saving, it can be associated with complications such as ventilator-induced lung injury and nosocomial pneumonia as recently nicely summarized by Newth et al (5). Endotracheal tubes (ETT) are uncomfortable for patients and increase the need for sedatives. An ETT in the upper airway can be associated with airway injury, particularly in mobile young patients. Furthermore, positive pressure ventilation may contribute to cardiovascular instability from heart-lung interactions. Therefore, it is important that MV be discontinued as soon as the patient is capable of sustaining spontaneous breathing. However, the experience in adults suggests that premature extubation may also be problematic and result in emergent reintubation with attendant complications, including the potential of catastrophic morbidity. A high mortality rate has been documented in both pediatric and adult patients who have required reintubation after extubation failure. Extubation failure is independently associated with a five-fold increased risk of death in pediatric patients. Consequently, although expeditious weaning and extubation are the goal, premature extubation can be lethal. Over 50% of ventilated PICU patients will have been extubated by 48 hrs after admission, but the rest often require prolonged ventilatory support. Both premature and delayed extubation increases morbidity and mortality as well as costs.

   Initiation of weaning and timing of extubation have been largely neglected in the pediatric literature (5). Weaning is the transition from ventilatory support to completely spontaneous breathing, during which time the patient assumes the responsibility for effective gas exchange while positive pressure support is withdrawn. There is no standard method of weaning. Indeed, there is disagreement about when the onset of weaning actually occurs and no validated, objective criteria as to when a patient can be extubated (6-9).

   The most common approach to weaning infants and children is gradual reduction of ventilatory support. Weaning with intermittent mandatory ventilation (IMV) or synchronized IMV (SIMV) occurs by reducing the ventilatory rate. With pressure support (PS) ventilation, the inspiratory pressure is initially set to provide the required support and then reduced gradually. PS is often combined with IMV/SIMV during weaning (SIMV-PS). Alternatively, another approach to weaning is attempted with alternating periods of complete ventilatory support and graded spontaneous breathing with assistance. This "sprinting" is performed on the theory that the respiratory muscles can be slowly trained to sustain complete spontaneous breathing. Also, theoretically this "sprinting" allows a better distribution of the tidal volume in the lung. Interestingly, both approaches are used simultaneously: the decision to use either one or both approaches is dependent upon the preferences of the attending physician as described in many observational single center studies.

   Importantly, there is no data comparing the "sprinting approach with more traditional approaches of weaning in children with respect to patient work-of-breathing. Work-of-breathing is defined by the physiologic work a patient has to deliver to expand the lungs and the chest wall. It can be assessed by various means:
   * Bedside: tachypnoea and the presence of nasal flaring and intercostal and/or interjugular retractions indicate increased work of breathing
   * Clinical surrogate parameters: the ratio of the inspiratory time to total breathing cycle time, the oesophageal pressure - rate product (PRP), oesophageal pressure - time product (PTP) and expiratory airway resistance (i.e. the difference in transpulmonary pressure and compliance, divided by flow). These clinical surrogate parameters require the presence of an oeosphageal catheter to measure the pressure. These catheters are routinely present in ventilated patients as they are used for nasogastric tube feeding; modern catheters can also measure the oesophageal pressure (i.e. double function).
   * Mathematically: the area under the oesophageal pressure - volume curve. This is the classic and traditional approach to measure work of breathing. Its normal value is within the range of 0.5 - 1.0 J/L. The variable is measured by a commercially available ventilator (AVEA, CareFusion, Yorba Linda, CA, USA). To measure this parameter, an oesophageal catheter is necessary.

   Children ventilated in the PICU of the Beatrix Children's Hospital are weaned from the mechanical ventilator using both the gradual weaning and the sprinting approach. In practice, this means that the patient is assessed by the attending physician on a daily basis if he or she can be weaned off the ventilator. If so, the ventilator mode is switched to PS ventilation (step 1). The level of PS is set to meet the level of PS set when the patient is ventilated in the SIMV-PS mode. The patient will be in the PS mode until he or she clinically shows increased work-of-breathing (tachypnoea and the presence of nasal flaring and intercostal and/or interjugular retractions indicate increased work of breathing). Then the patient is switched back to SIMV-PS but with a lower rate of breaths per minute delivered by the ventilator, allowing for more spontaneous breaths (step 2). The patient will be in this mode until he or she clinically shows increased work-of-breathing. If so, then the patient is switched back to full SIMV-PS.

   For this research proposal, we want to daily measure the work-of-breathing using the clinical surrogate parameters (PRP and PTP) and the traditional approach (the area under the oesophageal pressure - volume curve) when the patient is weaned off the ventilator. There will be no intervention, and the decision to wean the patient is left at the discretion of the attending physician. Ultimately, a better understanding of the work-of-breathing during weaning will help in the design of weaning protocols.
2. OBJECTIVES The primary objective for this study is to compare the level and time course for each patient of the work-of-breathing during PS ventilation (step 1) with the work-of-breathing during SIMV-PS ventilation with a lower rate of breaths per minute delivered by the ventilator (step 2).

   The secondary objectives for this study are to compare the level and time course of the PRP, PTP, and the PaO2/FiO2 ratio as well as the distribution of tidal volume in the lung during PS ventilation (step 1) with the work-of-breathing during SIMV-PS ventilation with a lower rate of breaths per minute delivered by the ventilator (step 2).
3. STUDY DESIGN This is a prospective exploratory study without invasive measurements in a 20 bed tertiary paediatric intensive care facility at the Beatrix Children's Hospital/University Medical Centre Groningen. The study will start December 1, 2011 and is completed by November 30, 2012.
4. STUDY POPULATION 4.1 Population (base) All mechanically ventilated children aged 0 to 5 years with or without lung pathology admitted to the paediatric intensive care unit are eligible for inclusion. Our PICU annually admits approximately 800 - 900 patients; nearly half of them require mechanical ventilation of which approximately 25% is ventilated for at least 24 hours. Thus, approximately 200 - 225 patients are annually eligible.

   4.2 Inclusion criteria
   * mechanical ventilation for at least 48 hours before the start of weaning
   * weight ≥ 3 kg
   * deemed eligible for weaning by the attending physician
   * stable haemodynamics, defined by the absence of need for increase in vaso-active drugs and/or fluid challenges at least 6 hours prior to enrolment 4.3 Exclusion criteria
   * mechanical ventilation less than 48 hours for unplanned admissions before the start of weaning
   * post-operative admission with expected duration of mechanical ventilaton less than 48 hours
   * not eligible for weaning as assessed by the attending physician (usually when there are unstable ventilator settings, defined by the need for increase of inspiratory pressures or positive end-expiratory pressure, and a FiO2 > 0.6 within 6 hours prior to enrolment)
   * unstable haemodynamics, defined by the need for increase in vaso-active drugs and/or fluid challenges within 6 hours prior to enrolment
   * admitted to the neonatal intensive care unit
   * premature birth with gestational age corrected for post-conceptional age less than 40 weeks
   * congenital or acquired neuromuscular disorders
   * congenital or acquired central nervous system disorders with depressed respiratory drive
   * severe traumatic brain injury (i.e. Glasgow Coma Scale < 8)
   * congenital or acquired damage to the phrenic nerve
   * congenital or acquired paralysis of the diaphragm
   * use of neuromuscular blockade prior to enrolment
   * uncorrected congenital heart disorder
   * chronic lung disease
   * severe pulmonary hypertension 4.4 Sample size calculation This study is designed to measure the differences over time in work-of-breathing within each patient at two different conditions (as outlined above, step 1 and step 2). To detect a difference of 0.2 J/L in work of breathing measured by the area under the pressure-volume curve (expressed in J/L) between step 1 and step 2, we need a sample size of 24 patients to study an actual effect standard deviation of 0.25 J/L with 80% power and 5% significance. We aim to study patients with and without lung injury. Therefore, patients will be categorized as having lung injury defined as Acute Hypoxaemic Respiratory Failure (AHRF) or no lung injury. AHRF is defined as a) the presence of one or more (bilateral) abormalities on chest radiograph, b) PaO2/FiO2 ratio < 300 mmHg and c) acute onset.

   Thus, a total sample size of 48 (N = 24 with AHRF and N = 24 without AHRF) is required.
5. METHODS 5.1 Study parameters/endpoints 5.1.1 Main study parameter/endpoint The level and time course of the patient work-of-breathing measured by the area under the pressure-volume curve during PS ventilation (step 1) with the work-of-breathing during SIMV-PS ventilation with a lower rate of breaths per minute delivered by the ventilator (step 2).

   5.1.2 Secondary study parameters/endpoints
   * The level and time course of the clinical surrogate parameters for work-of-breathing:
   * Oesophageal pressure - time product (PTP)
   * Oesophageal pressure - rate product (PRP)
   * Expiratory airway resistance
   * Distribution of tidal volume during PS ventilation (step 1) compared with SIMV-PS ventilation with a lower rate of breaths per minute delivered by the ventilator (step 2)
   * The level and time course of oxygenation as defined by the PaO2/FiO2 ratio during PS ventilation (step 1) with the work-of-breathing during SIMV-PS ventilation with a lower rate of breaths per minute delivered by the ventilator (step 2)

   5.2 Study procedures Standard care All children are put on a time-cycled, pressure limited ventilation mode (AVEA, CareFusion, Yorba Linda, CA, USA). Inspiratory pressures are set to deliver a expiratory tidal volume of 4- 12 ml/kg ideal bodyweight. The frequency of the delivered machine-breaths is set in accordance with age and disease condition of the patient. All patients have an indwelling arterial catheter for blood sampling and haemodynamic measurements. Enteral feeding is ensured through a nasogastric tube. This nasogastric tube is also capable of measuring the oesophageal pressure via a small balloon that needs to be inflated with less than 2 mL of water. The correct position is confirmed by the nurse taking care of the patient in accordance with local nursing guidelines; to evaluate if the small balloon is positioned correctly, the oesophageal flow - time curve is observed for the presence of the cardiac signal. Mild sedation is achieved using benzodiazepines (either through continuous intravenous infusion or intermittent administration) and opiates. Blood samples (0.5 mL) are routinely drawn 6 times a day for measuring the PaCO2 and PaO2.

   Before start of the study the patient will be assessed if he or she is able to initiate and maintain spontaneous breathing.

   Children ventilated in the PICU of the Beatrix Children's Hospital are weaned from the mechanical ventilator using both the gradual weaning and the sprinting approach. In practice, this means that the patient is assessed by the attending physician on a daily basis if he or she can be weaned off the ventilator. If so, the ventilator mode is switched to PS ventilation (step 1). The level of PS is set to meet the level of PS set when the patient is ventilated in the SIMV-PS mode. The patient will be in the PS mode until he or she clinically shows increased work-of-breathing (tachypnoea and the presence of nasal flaring and intercostal and/or interjugular retractions indicate increased work of breathing). Then the patient is switched back to SIMV-PS but with a lower rate of breaths per minute delivered by the ventilator, allowing for more spontaneous breaths (step 2). The patient will be in this mode until he or she clinically shows increased work-of-breathing. If so, then the patient is switched back to full SIMV-PS. Of note, the time lap between step 1 and step 2 increases when the child clinically improves.

   There will be no intervention, and the decision to wean the patient is left at the discretion of the attending physician.

   Study protocol Collection of clinical data from the patient's medical chart. Clinical data include PIM II and PRISM III score, demographical data including gender, age and weight, and admission diagnosis. Ventilation parameters measured by the mechanical ventilation (including level of positive inspiratory pressure, level of positive end-expiratory pressure, inspiration time, and expiratory tidal volume) and the PaO2/FiO2 are recorded on a daily basis. The PaO2/FiO2 ratio is calculated by dividing the arterial PaO2 by the administered FiO2, the oxygenation index is calculated as follows: mean airway pressure * FiO2* 100 divided by the PaO2. A small blood sample (0.5 mL) is drawn from the already routinely present indwelling peripheral arterial line to measure the PaO2 and PaCO2.

   Measurements for work-of-breathing Respiratory system mechanics are measured using a pneumotachograph/pressure transducer system available in the ventilator (Bicore II, CareFusion, Yorba Linda, CA, USA). Airway pressure (Paw) and flow (V) are measured at the proximal end of the endotracheal tube. Tidal volume (Vt) and minute ventilation are obtained by integrating the flow signal. From the flow signal, the respiratory frequency, inspiratory time (Ti) and total respiratory cycle duration (Ttot) are measured. The duty cycle, defined by Ti/Ttot, and mean inspiratory flow are calculated.

   Figure 1 Airway pressure (Pao), flow (inspiration upward), and esophageal pressure (Pes) tracings. The hatched area represents integration of the Pes versus either time or volume. The dotted area shows contribution of the chest wall recoil pressure to pressure-time product or work of breathing.

   Work of breathing is assessed by measuring the area enclosed between the oesophageal pressure-volume loop during inspiration and the relaxation curve of the chest wall using the Campbell technique (Figure 1). The work of breathing is evaluated per breath during each respiratory cycle and expressed as J*min-1*kg bodyweight. The negative deflection of oesophageal pressure during inspiration (ΔPes) is calculated as the difference between the end-expiratory oesophageal pressure and the lowest oesophageal pressure. ΔPes represents the inspiratory work of breathing. The pressure-time product (PTP) is calculated as the area subtended by the Pes tracing and the chest wall static recoil pressure for inspiratory time (Figure 1). PTP is expressed as cmH2O*s*min-1. The pressure-rate product (PRP) is calculated by mean change in oesophageal pressure times the respiratory rate. Work of breathing is displayed by the ventilator, PTP and PRP and displayed by a WOB and paediatric mechanical ventilation separate pulmonary function monitor connected to the ventilator (BiCore II, CareFusion, Yorba Linda, CA, USA).

   Measurements for distribution of tidal volume The distribution of tidal volume will be measured by electrical impedance tomography (EIT) using the Göttingen Goe-MF II EIT system (CareFusion, Yorba Linda, CA, USA). Sixteen electrodes (Blue Sensor BR(S)-50-K, Ambu, Denmark) are applied circumferentially around the infant's chest at the mammary line for EIT measurements. All measurements are made at a scan rate of 48 Hz for 60 seconds. A 5 mA peak-to-peak, 50 kHz electrical current will be injected at each adjacent electrode pair and the resultant potential differences are measured at the remaining adjacent electrode pairs. Subsequently, all adjacent electrode pairs are used for current injection, thus completing one data cycle. The impedance map will be built using the back-projection image reconstruction algorithm. It calculates the relative impedance ΔZ, defined by [Zinst - Zref] / Zref (where Zinst is the instantaneous local impedance and Zref the reference impedance, determined from each cycle of current injections and voltage measurements in each pixel). Both the respiratory and cardiac components of the EIT signal are identified in the frequency spectra generated from all EIT measurements (Fourier transformation). Cut-off frequency of the low-pass filter will be set below the heart rate (0.67 Hz, 40 beats/min) to eliminate the cardiac signal from the impedance measurements. The calculations performed on the sums of values from all pixels of the 32 x 32 pixel matrix EIT image are described as "global". In addition, sums of values from the left and right lung regions are described separately, and the entire EIT image will be divided into 64 regions-of-interest (ROI) (32 left and 32 right lung) from anterior to posterior as previously described by Frerichs and co-workers. Ventilation-induced tidal volume (ΔZVt) will be quantified by measuring the relative ΔZ from the highest point at end inspiration to the lowest point at end expiration, and an average ΔZ will be calculated from multiple breaths. Changes in ΔZVt were calibrated to volume using the known Vt. End-expiratory lung volume will be determined by measuring the median impedance from the lowest point at expiration during the sampling time (ZEELV), that is calibrated to volume (EELV) using the known VT and ΔZVT.

   All of the outlined measurements will be made once a day during the weaning process.

   5.3 Withdrawal of individual subjects All patients will remain in the study as there is no interference with clinical practice (unless parents or legal caretakers withdraw their consent). As discussed, the patient is clinically assessed between the two weaning approaches for clinical signs of increased work-of-breathing. The patient will be in the PS mode until he or she clinically shows increased work-of-breathing (tachypnoea and the presence of nasal flaring and intercostal and/or interjugular retractions indicate increased work of breathing). Then the patient is switched back to SIMV-PS but with a lower rate of breaths per minute delivered by the ventilator, allowing for more spontaneous breaths. The patient will be in this mode until he or she clinically shows increased work-of-breathing. If so, then the patient is switched back to full SIMV-PS.
6. SAFETY REPORTING 6.1 Section 10 WMO event In accordance to section 10, subsection 1, of the WMO, the investigator will inform the subjects and the reviewing accredited METC if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal. The study will be suspended pending further review by the accredited METC, except insofar as suspension would jeopardise the subjects' health. The investigator will take care that all subjects are kept informed.

   6.2 Adverse and serious adverse events Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the experimental treatment. All adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded.

   A serious adverse event is any untoward medical occurrence or effect that at any dose:
   * results in death;
   * is life threatening (at the time of the event);
   * requires hospitalisation or prolongation of existing inpatients' hospitalisation;
   * results in persistent or significant disability or incapacity;
   * is a congenital anomaly or birth defect;
   * is a new event of the trial likely to affect the safety of the subjects, such as an unexpected outcome of an adverse reaction, lack of efficacy of an IMP used for the treatment of a life threatening disease, major safety finding from a newly completed animal study, etc.

   All SAEs will be reported through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 15 days after the sponsor has first knowledge of the serious adverse reactions. SAEs that result in death or are life threatening should be reported expedited. The expedited reporting will occur not later than 7 days after the responsible investigator has first knowledge of the adverse reaction. This is for a preliminary report with another 8 days for completion of the report.

   6.2.1 Annual safety report In addition to the expedited reporting of SUSARs, the sponsor will submit, once a year throughout the clinical trial, a safety report to the accredited METC, competent authority, Medicine Evaluation Board and competent authorities of the concerned Member States.

   This safety report consists of:
   * a list of all suspected (unexpected or expected) serious adverse reactions, along with an aggregated summary table of all reported serious adverse reactions, ordered by organ system, per study
   * a report concerning the safety of the subjects, consisting of a complete safety analysis and an evaluation of the balance between the efficacy and the harmfulness of the medicine under investigation.

   6.3 Follow-up of adverse events All adverse events will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist.
7. STATISTICAL ANALYSIS 7.1 Descriptive statistics At first, continuous data will be examined if they display a normal distribution. If so, then these data are presented as presented as mean ± standard deviation. The continuous data that do not show a normal distribution are presented as median + 25-75% interquartile range (IQR). Dichotomous data or categorical data is presented as percentage of total. Patients will be categorized according to the presence or absence of lung injury.

7.2 Univariate analysis The collected clinical data (i.e. demographics, severity of illness, admission diagnosis etc) is used to characterize the study population.

Primary outcome measure: the work-of-breathing measured by the area under the pressure-volume curve will be analyzed using either the paired t -test or the Wilcoxon signed rank test (depending on the distribution of the variable) between baseline and step 1, and between step 1 and step 2. Separate analyses will be performed for patients with and without lung injury.

Secondary outcome measure: the oesophageal pressure - time (PTP) and oesophageal pressure - rate product (PRP), and the PaO2/FiO2 ratio will also be analyzed using the paired t -test or the Wilcoxon signed rank test (depending on the distribution of the variable) between baseline and step 1, and between step 1 and step 2 as outlined above. The distribution of the tidal volume is expressed as a ratio between 0 and 1 (with 0 being ventral ventilation and 1 being dorsal ventilation). Hence, this ratio will also be analyzed using the paired t -test or the Wilcoxon signed rank test (depending on the distribution of the variable) between baseline and step 1, and between step 1 and step 2 as outlined above. Also, separate analyses will be performed for patients with and without lung injury.

All analyses are performed using SPSS for MacIntosh v18 (Chicago, Ill, USA). P < 0.05 is accepted as statistically significant.

Stopping rule: the patient is clinically assessed between the two weaning approaches for clinical signs of increased work-of-breathing. The patient will be in the PS mode until he or she clinically shows increased work-of-breathing (tachypnoea and the presence of nasal flaring and intercostal and/or interjugular retractions indicate increased work of breathing). Then the patient is switched back to SIMV-PS but with a lower rate of breaths per minute delivered by the ventilator, allowing for more spontaneous breaths. The patient will be in this mode until he or she clinically shows increased work-of-breathing. If so, then the patient is switched back to full SIMV-PS.

ELIGIBILITY:
Inclusion Criteria:

* aged 0 to 5 years with or without lung pathology admitted to the paediatric intensive care unit are eligible for inclusion
* mechanical ventilation for at least 48 hours before the start of weaning
* weight ≥ 3 kg
* deemed eligible for weaning by the attending physician, i.e. able to initiate and maintain spontaneous breathing.
* stable haemodynamics, defined by the absence of need for increase in vaso-active drugs and/or fluid challenges at least 6 hours prior to enrolment

Exclusion Criteria:

* mechanical ventilation less than 48 hours for unplanned admissions before the start of weaning
* post-operative admission with expected duration of mechanical ventilaton less than 48 hours
* not eligible for weaning as assessed by the attending physician (usually when there are unstable ventilator settings, defined by the need for increase of inspiratory pressures or positive end-expiratory pressure, and a FiO2 > 0.6 within 6 hours prior to enrolment)
* unstable haemodynamics, defined by the need for increase in vaso-active drugs and/or fluid challenges within 6 hours prior to enrolment
* admitted to the neonatal intensive care unit
* premature birth with gestational age corrected for post-conceptional age less than 40 weeks
* congenital or acquired neuromuscular disorders
* congenital or acquired central nervous system disorders with depressed respiratory drive
* severe traumatic brain injury (i.e. Glasgow Coma Scale < 8)
* congenital or acquired damage to the phrenic nerve
* congenital or acquired paralysis of the diaphragm
* use of neuromuscular blockade prior to enrolment
* uncorrected congenital heart disorder
* chronic lung disease
* severe pulmonary hypertension

Ages: 0 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
The work of breathing (Campbell Diagram) | 10 minutes
  The level and time course of the patient work-of-breathing measured by the area under the pressure-volume curve during PS ventilation with the work-of-breathing during SIMV-PS ventilation with a lower rate of breaths per minute delivered by the ventilator.

SECONDARY OUTCOMES:
Pressure-time-product (PTP) | 10 minutes
  Calculated by the integral of the esophageal signal over time during inspiration multiplied by respiratory rate
Pressure-rate-product (PRP) | 10 minutes
  The difference between the peak esophageal pressure and bottom esophageal pressure during one inspiration multiplied by the respiratory rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Beatrix Children's Hospital, University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koopman AA, van Dijk J, Oppersma E, Blokpoel RGT, Kneyber MCJ. Surface electromyography to quantify neuro-respiratory drive and neuro-mechanical coupling in mechanically ventilated children. Respir Res. 2023 Mar 13;24(1):77. doi: 10.1186/s12931-023-02374-w. PMID 36915106
- [Derived] van Dijk J, Koopman AA, de Langen LB, Dijkstra S, Burgerhof JGM, Blokpoel RGT, Kneyber MCJ. Effect of pediatric ventilation weaning technique on work of breathing. Respir Res. 2022 Jul 13;23(1):184. doi: 10.1186/s12931-022-02106-6. PMID 35831900